CLINICAL TRIAL: NCT05569642
Title: A Study of Cluster Analysis to Identify Metabolic Syndrome Components and Physical Fitness in Patients With Metabolic Syndrome
Brief Title: Cluster Analysis to Identify Metabolic Syndrome Components and Physical Fitness in Patients With Metabolic Syndrome
Status: Completed | Type: Observational
Sponsor: Istanbul Galata University (Other)
Responsible Party: Sponsor
Other Study IDs: IstanbulGalataUni
Record Dates: First submitted 2022-09-24; First posted 2022-10-06 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2022-06

CONDITIONS: Metabolic Syndrome
Keywords: MetS, physical fitness, physical activity, cluster analysis
MeSH Terms: conditions — Metabolic Syndrome; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The components of MetS (abdominal obesity, high blood pressure, high serum glucose, high triglyceride level and low HDL-C) differ according to demographic characteristics such as age, gender and comorbidities. Low physical activity level, genetic makeup, nutritional disorders, decreased muscle strength and low cardiorespiratory fitness can be counted among the risk factors associated with MetS. In our study, it was aimed to examine the relationship between the components of the MetS and muscle strength, physical activity, functional capacity and quality of life. Our secondary aim is to investigate the independent effects of different components of MetS on each parameter.

DETAILED DESCRIPTION:
The participants' sociodemographic characteristics such as age, height, weight, body mass index, waist circumference, marital status and education level, and anthropometric measurements, body fat percentage distributions, fasting blood glucose, HbA1c and lipid profiles will be recorded from previous analysis reports. Lower extremity quadriceps muscle strength Hand-held dynamometer, grip strength hand dynamometer, physical activity level International Physical Activity Questionnaire-Short Form-IPAQ-SF, number of steps pedometer, functional capacity 6 minute walking test and quality of life will be evaluated with the European Quality of Life Scale-5 Dimension.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed with MetS by an Internal Medicine Specialist according to NCEP-ATP III criteria
* Finding abdominal obesity component according to TURDEP-II criteria
* Being between the ages of 40-65
* To be able to read and write Turkish
* Having signed the informed consent form

Exclusion Criteria:

* Lack of cooperation
* Those with severe peripheral or central neurological disorders
* Patients with uncontrolled hypertension and uncontrolled arrhythmia
* Pregnant or breastfeeding patients
* Those with diabetic ulcer or neuropathy
* Chronic kidney failure (eGFR<30 ml/min)
* Chronic liver disease (ALT/AST<3X Normal upper limit)
* Those with serious respiratory system disease
* Patients with cardiac pacemaker
* History of previous stroke or myocardial infarction
* Presence of lower and upper extremity orthopedic problems that may prevent the application of clinical tests

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteers between the ages of 40-65, who have been diagnosed with MetS on the basis of type 2 diabetes for at least one year by an Internal Medicine Specialist, applying to the Department of Endocrinology and Metabolism Diseases, Department of Internal Medicine, Istanbul University, Istanbul Medical Faculty, will be included in the study.
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Measurement of Lower Extremity Muscle Strength | 7 minutes.
  Measurement of Lower Extremity Muscle Strength: A hand-held dynamometer will be used to evaluate quadriceps muscle strength. While the individual is in the sitting position, the arms will be crossed over the chest and the hips and knees will be flexed to 90º. Then, the individual will be asked to bring the knee to full extension and make a maximal voluntary contraction for 5 seconds against the resistance applied by the dynamometer placed on the distal part of the leg. The average value will be recorded in kg/Newton.
The 6-minute walking test (6MWT) | 6 minutes.
  Functional Capacity Measurement: The 6-minute walking test (6MWT) will be used to evaluate the functional exercise capacity of individuals. The 6MWT is a valid and reliable test, easy to administer, well tolerated, and more reflective of activities of daily living than other tests. The test will be applied according to the criteria of the American Thoracic Society (ATS). Patients will rest for at least 10 minutes before the test. They will then be asked to walk as fast as they can but without running in 6 minutes on a straight 30-meter corridor. During the test they will be encouraged to walk fast using their maximum speed. Oxygen saturation and heart rates of the patients before and after the test will be evaluated with Baseline® finger pulse oximeter, systolic and diastolic blood pressures with sphygmomanometer, dyspnea and fatigue levels will be evaluated with Modified Borg Scale. At the end of the test, the distance that patients can walk (6MWM) will be recorded in meters.
Physical activity levels of individuals will be determined by IPAQ-SF scale | 8 minutes.
  Physical activity levels of individuals will be determined by IPAQ-SF. In the study, the self-administered short form of the questionnaire, which includes "the last seven days", will be used to evaluate the level of physical activity. This short form consists of seven questions and provides information about sitting, walking, moderate-intensity activities, and time spent in vigorous activities. In addition, there is a sitting question to determine the sedentary time. However, it is not included in the scoring. Calculation of the total score of the short form includes the sum of time (minutes) and frequency (days) of walking, moderate-intensity activity, and vigorous activity. In the evaluation of all activities, the criterion is that each activity is done for at least 10 minutes at a time.
Measurement of step counts by Pedometers | The participant's step count will be tracked for 7 days.
  Step Count Measurement: Pedometers (pedometers); It is a portable, easy-to-use tool that can objectively measure the number of steps, kilometers walked, and is used to evaluate the level of daily physical activity. It is a sensor sensitive to mechanical movement during walking. Pedometers have been shown to be the most valid method for evaluating step counts. The individuals participating in our study will be introduced to the OMRON branded Walking style One 2.1 pedometer device, validated by De Craemer et al., and will be taught to use it. Then, individuals will be asked to carry this pedometer all day for a week, in the waist area or in the pocket. The pedometer used has the feature of recording the number of steps, energy expenditure level (kcal) and the time spent with active movement with its 3D sensor, 7-day retrospective memory. After one week of use, the data recorded with the pedometer will be taken.
Grip Strength Measurement | 5 minutes.
  Grip Strength Measurement: A Jamar brand hydraulic type dynamometer will be used to measure the grip strength of the participants. It will be performed with the individual in a sitting position on an unsupported chair, shoulder adduction, elbow 90º flexion, forearm in neutral position, wrist in 0-30° extension and 0-15° ulnar deviation. Participants will be asked to squeeze the dynamometer with maximum effort for 5 seconds with their dominant hand and then leave it completely relaxed. The average of the obtained values will be recorded in "pounds".

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine, Department of Internal Medicine, Department of Endocrinology and Metabolic Diseases, Istanbul, Turkey (Türkiye)